CLINICAL TRIAL: NCT06613971
Title: Dynamic Light Scattering Ocular Measurement in the Detection of Dementia
Acronym: DLS
Status: Recruiting | Type: Observational
Sponsor: MD Stem Cells (Industry)
Collaborators: Jeffrey N Weiss MD (Unknown); 3T Radiology (Unknown); The Healing Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: ACRM2024003
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2024-09

CONDITIONS: Dementia; Dementia Alzheimer Type
Keywords: Dementia; Spectroscopy; Dynamic Light Scattering Spectroscopy; Retinal Nerve Fiber Layer; DLS
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients diagnosed with dementia: Patients diagnosed with dementia including those caused by Alzheimer's, Vascular, Lewy body, Mixed, Parkinson's, Frontotemporal, Creutzfeldt-Jakob, Normal pressure hydrocephalus, Huntington's, Wernicke-Korsakoff Syndrome.
- Patients without cerebral pathology: Patients without cerebral pathology (no dementia)

SUMMARY:
This is a human clinical study making a noninvasive measurement from a patient's eye to determine whether there is a quantitative difference in measurements between patients with and without the diagnosis of dementia.

DETAILED DESCRIPTION:
1. Type of Research

   This is a human clinical study making a noninvasive measurement from a patient's eye to determine whether there is a quantitative difference in measurements between patients with and without the diagnosis of dementia.

   This research is not federally funded nor subject to federal oversight.
2. Purpose and Objective of the Study

   The purpose of the study is to determine whether dynamic light scattering spectroscopy, also known as laser light scattering spectroscopy, or photon correlation spectroscopy, a noninvasive quantitative technique, has utility in the diagnosis of dementia. The objective is to determine which types of dementia and at what stages they may be most effectively detected.
3. Background of the Study

Study Rationale

Dementia is a common cause of morbidity and mortality. It is caused by physical changes in the brain that causes the loss of mental abilities and memory that affect the activities of daily living. The types of dementia include: Alzheimer's disease, Vascular dementia, Dementia with Lewy bodies, Mixed dementia, Parkinson's disease, Frontotemporal dementia, Creutzfeldt-Jakob disease, Normal pressure hydrocephalus, Huntington's disease, Wernicke-Korsakoff Syndrome, etc.

Alzheimer's disease is a slowly progressive brain disease beginning prior to the appearance of symptoms and accounts for approximately 60 - 80% of dementia cases. Definitive diagnosis is made posthumously with the discovery of protein fragment beta-amyloid plaques and twisted strands of the protein tau (tangles) with nerve cell damage and death.

Vascular dementia, previously known as post-stroke or multi-infarct dementia is solely diagnosed in approximately 10% of dementia cases. The development of Lewy bodies in the cerebral cortex can cause dementia. The type of aggregate pattern may be indicative of Dementia with Lewy bodies or of Parkinson's disease.

Abnormalities of more than one dementia cause may occur simultaneously in the brain causing a mixed dementia. In Parkinson's disease, the alpha-synuclein clumps generally occur in a deep area of the brain called the substantia nigra and are thought to affect the production of dopamine.

In Normal Pressure Hydrocephalus an abnormal increase of fluid in the brain leads to dementia. This may sometimes be corrected by the placement of a shunt in the brain to drain the excess fluid. There are no definite distinguishing microscopic abnormalities seen in all cases of frontotemporal dementia.

Creutzfeldt-Jakob disease (mad-cow disease) is caused by an infection with a prion. Huntington's disease is caused by a defective gene on chromosome 4. Vitamin B-1 deficiency (thiamine), generally caused by alcoholism, is the cause of Wernicke-Korsakoff syndrome.

In the absence of dementia etiology, as seen in Creutzfeldt-Jakob disease, Normal Pressure Hydrocephalus, Huntington's disease, Wernicke-Korsakoff syndrome, the true diagnosis is generally made pathologically, after the patient has expired.

During the last 15 years there have been more than 500 clinical trials of therapeutic agents for Alzheimer's disease registered with the National Institute of Health website, clinicaltrials.gov. For those trials with reported results, the failure rate has been almost 100%. Though most trials typically last 1.5 to 3 years, it has been estimated that, depending on the efficacy of the therapeutic intervention, study duration would need to be 5 - 10 years in duration to detect an effect.

Therefore, what is needed is a sensitive, quantitative, technique that can detect the beginnings or early onset of these conditions before the development of symptoms.

The retina is visible within the eye and is composed of 10 histologic layers. The nerve fiber layer of the retina is an extension of the brain. The early detection of neurologic damage at the microscopic level when it is still potentially reversible is a prerequisite for the development of potential cures. The early detection of the effectiveness of treatment allows for better and more effective treatments.

It has been demonstrated that patients with Alzheimer's disease have thinning of the retinal nerve fiber layer and retinal ganglion cell layer by ocular coherence tomography (OCT) images and measurements taken through the macula and peripapillary areas. This is consistent with histopathologic data. Inner retina thinning has been correlated with disease severity. This may be related to the presence of amyloid-beta within the retina.

Inner retinal thinning has been found in other neurodegenerative diseases including multiple sclerosis, amyotrophic lateral sclerosis, dementia with Lewy bodies, and multiple system atrophy.

As compared to the inner retinal thinning seen in Alzheimer's disease, thinning of the photoreceptor or outer retina thinning has been found in frontotemporal degeneration. Approximately 30% of patients initially diagnosed with frontotemporal degeneration are subsequently diagnosed with Alzheimer's disease at autopsy.

Dynamic Light Scattering (DLS) measures the scattered light intensity fluctuations resulting from thermal random motion (Brownian motion). It has been used to predict the development of cataracts in rabbits, and detect the development of cataract formation and of diabetes mellitus in humans. The results demonstrated the utility of DLS to noninvasively quantitate subtle changes at the molecular level.

A proof-of-concept instrument for making retinal measurements has been developed. The system provides optical power below the maximal permissible exposure recommended by the ANSI Z136.1 standard. The minimal amount of light necessary to make a 5 second measurement is used. The detection system is interfaced with a standard clinical fundus camera. The intensity fluctuations are averaged over 5 seconds and the cumulant analysis method used to analyze the resulting autocorrelation function.

17 patients were tested using this device and no significant difference was seen between the left and the right eye in patients with normal eye examinations. In addition, the results, taken over a 6-month time span were not significantly different, demonstrating reproducibility.

The ability to quantitatively and objectively detect molecular changes, before they become observable by standard imaging techniques allows the early detection and monitoring of patients with conditions affecting the retina, such as dementia.

Appendix A

DLS publications

4. Participant Selection

A. Inclusion and Exclusion Criteria

Inclusion:

To be eligible for the study patients must:

1. Have either a documented diagnosis of dementia or no neurologic condition of cerebral origin.
2. Have no ophthalmic history of pathology, except for refractive error or cataract.
3. Be over the age of 18.
4. Be medically stable.

Restrictions:

1. All patients must be capable of an adequate ophthalmic evaluation and testing. This includes the ability to cooperate with the exam, sufficiently clear media (cornea, lens, vitreous) and sufficient pupillary dilation.
2. Patients must be capable of providing informed consent.
3. Patients who are not medically stable or who may be at significant risk to their health will not be eligible.
4. Women of child bearing age must not be pregnant at the time of examination.

   B. Gender - no restrictions. Women of child bearing age are eligible but must not be pregnant at the time of treatment.

   C. Racial/ Ethnic origin- no restrictions.

   D. Vulnerable populations - no vulnerable populations will be eligible.

   E. Age- no patients under the age of 18 are to be enrolled. For those 18 years and older there will be no age restrictions.

   F. Total number of Participants to be Enrolled: 50 25 patients diagnosed with dementia 25 age-matched patients without cerebral pathology
5. STUDY DESIGN / METHOD / PROCEDURES A. Summary of Research Design

   This is an office-based study. Patients referred by Dr. Eber, or associates, for study inclusion will be interviewed. An ophthalmic history will be taken. If the patient is eligible for study participation, they will undergo pharmacologic dilation of one eye. The dilated eye will be chosen by the patient. Standard ophthalmic drops used for mydriasis will be utilized. After approximately 10 - 15 minutes, a DLS measurement will be performed. It is estimated that the entire test will take 5 minutes to complete. The patient will be instructed that the dilation will wear off in approximately 2 - 3 hours.

   B. Performance of Measurements

   Dynamic Light Scattering (DLS) Device - The patient fixates with their undilated eye at an external light. A standard, commercially available fundus camera is focused on the retina. The DLS light is parfocal with the fundus camera. The DLS operator (Dr. Weiss) presses a button and a 5 second duration measurement is made.

   C. General Side Effects

   The procedure includes the administration of standard ophthalmic medications to dilate the pupil. There is a very small chance that this may lead to an angle closure glaucoma. This is unlikely and has not been seen in Dr. Weiss' more than 30-year career as an ophthalmologist.

   D. Collection and used of data:

   Patients give permission for use of their medical information for their own care and for any publication, presentation or public communication about the procedure and results. In the case of non-direct patient care communication, the patient's name and contact information will be held in confidence and not released to protect privacy. However, if required by law, state or federal agencies may be given access to the full name, data, medical records and information. Access will be granted to the Institutional Review Board as they require for monitoring the study.
6. Analysis of Study Results Data will be collected and analyzed for significance. Standard statistical methodology will be used.

   A. Storage of Data Data will be stored in paper files and will be accessible by Dr. Weiss, his staff and associates. This will be kept in the usual manner as other medical files and for the required period of time by law.

   B. Confidentiality of Data All data will be maintained in a confidential manner equal to other medical data and records.
7. Risk/Benefit Assessment Risk and discomforts are considered "Minimal Risk". Pupillary dilation is a normal part of standard eye examination. The measurement light is much weaker than those lights used in a standard eye examination.

   A. Adverse Events Any Adverse Events (AE) or Serious Adverse Events (SAE) will be managed by Dr. Weiss at the time of the event. An Adverse Event will be defined as an event related to the procedure that has a high risk to cause permanent loss of vision or health to the patient. These will be reported to the IRB within 60 days of documentation. A Serious Adverse Event is defined as the permanent loss of vision or a permanent medical injury to the patient as a result of the procedure and will be reported to IRB within 45 business days of their documentation.

   B. Benefits Patients participating in this study will receive no direct benefits other than possibly helping to diagnose other patients with dementia.
8. Participant Recruitment and Informed Consent A. Recruiting Recruiting will be brought to the attention of potential patients through announcements made by Dr. Eber's office. Recruiting will continue until 50 patients have been enrolled. No coercion will be used. In the course of providing information about the study, it will be communicated that patients will be participating in a clinical study conducted under an IRB approved protocol.

B. Length of Study The study will begin on the date of IRB approval and continue until 50 patients are recruited for the study.

C. Informed Consent / Assent See Informed Consent

Appendix A

1. Weiss JN. Laser light scattering of in-vivo human lenses. Am J. Ophthalmol. (Letter to the Editor) 1982; 94:683.
2. Weiss JN. Laser device seen as aid to early detection of cataracts. Ophthalmol Times. (Interview) 1982; December 1:1.
3. Weiss JN. New laser technique detects eye disease, Joslin Diabetes Center newsletter. 1983; 11, 4:8.
4. Weiss JN, Rand LI, Gleason RE, Soeldner JS. Laser light scattering spectroscopy of in-vivo human lenses. Invest Ophthalmol Vis Sci. 1984; 25:594-598.
5. Nishio I, Weiss JN, Tanaka T, Clark JI, Giblin FJ, Reddy VN, Benedek GB. In-vivo observation of lens protein diffusivity in normal and X-irradiated rabbit lenses. Exp Eye Res. 1984; 39;61-68.
6. Bursell SE, Weiss JN, Eichold BH. Diagnostic Laser light scattering spectroscopy for human eyes. Proceedings of the International Congress on the Applications of Laser and Electro-optics. 1984; 43:61-67.
7. Weiss JN, Bursell SE, Gleason RE, Eichold BH. Photon correlation spectroscopy of in-vivo human cornea. Cornea. 5(1):19-24, 1986.
8. Bursell SE, Baker RS, Weiss JN, Haughton JF, Rand LI. Clinical photon correlation spectroscopy evaluation of human diabetic lenses. Exp. Eye Res. 49:241-58, 1989.
9. Bursell SE, Karalekas DP, Craig MS. The effect of acute changes in blood glucose on lenses in diabetic and non-diabetic subjects using quasi-elastic light scattering spectroscopy. Current Eye Research. 8:821-834, 1989. Bursell SE, Weiss JN, Karalekas DP, Craig MS. Correction Notice - Current Eye Research. 11(5):479, 1992.
10. Weiss JN, Letter to the Editor - DLS Technology Origins. Review of Ophthalmology. 16;12:11-12, 2009.
11. Weiss JN, Dynamic Light Scattering Technique Shows Potential in Measuring Effects of AMD Treatment. Ocular Surgery News, Retinal Edition. 31;8:57, 2013.
12. Weiss JN, Levy S. Dynamic Light Scattering Spectroscopy of the Retina - A non- invasive quantitative technique to objectively document visual improvement following ocular stem cell treatment. Stem Cell Investig. 2019;6:8 doi 10.21037/sci.2019.03.01.

ELIGIBILITY:
1. All patients must be capable of an adequate ophthalmic evaluation and testing. This includes the ability to cooperate with the exam, sufficiently clear media (cornea, lens, vitreous) and sufficient pupillary dilation.
2. Patients must be capable of providing informed consent.
3. Patients who are not medically stable or who may be at significant risk to their health will not be eligible.
4. Women of child bearing age must not be pregnant at the time of examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diagnostic radiology practice
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2027-04-25 (Estimated); Study Completion 2028-04-25 (Estimated)

PRIMARY OUTCOMES:
Comparison of Dynamic Light Scattering Spectroscopy in Dementias | Single measurement taken over 5 minutes
  Dynamic light scattering will be compared between patients with dementias and patients with no cerebral pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey N Weiss, MD, Principal Investigator — The Healing Institute
Locations (1):
- 3T Radiology, Coconut Creek, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
Uncertainty regarding how this would affect patient privacy. The Principal Investigator would need to understand exactly what was to be shared and if patient permission would be needed.